CLINICAL TRIAL: NCT01421121
Title: Safety and Immunogenicity of an Inactivated EV71 Vaccine in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EV71-1001-II
Record Dates: First submitted 2011-07-22; First posted 2011-08-22 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Infection, Viral, Enterovirus
MeSH Terms: conditions — Infections; Enterovirus Infections | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 100U EV71 vaccine with adjuvant (Experimental): 120 infants received 2 doses of 100U EV71 vaccine with aluminium hydroxide adjuvant 28 days apart
  Interventions: Biological: 100U EV71 vaccine with adjuvant
- 200 U EV71 vaccine with adjuvant (Experimental): 120 infants received 2 doses of 200U EV71 vaccine with aluminium hydroxide adjuvant 28 days apart
  Interventions: Biological: 200 U EV71 vaccine with adjuvant
- 400U EV71 vaccine with adjuvant (Experimental): 120 infants received 2 doses of 400U EV71 vaccine with aluminium hydroxide adjuvant 28 days apart
  Interventions: Biological: 400U EV71 vaccine with adjuvant
- 200U EV71 vaccine without adjuvant (Experimental): 60 infants received 2 doses of 200U EV71 vaccine without adjuvant 28 days apart
  Interventions: Biological: 200U EV71 vaccine without adjuvant
- Placebo (Placebo Comparator): 120 infants received 2 doses of placebo 28 days apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 100U EV71 vaccine with adjuvant — inactivated vaccine (vero cell) against EV71 of 100U /0.5ml, two doses, 28 days interval
  Other Names: EV71 vaccine
  Arms: 100U EV71 vaccine with adjuvant
Biological: 200 U EV71 vaccine with adjuvant — inactivated vaccine (vero cell) against EV71 of 200U /0.5ml, two doses, 28 days interval
  Other Names: EV71 vaccine
  Arms: 200 U EV71 vaccine with adjuvant
Biological: 400U EV71 vaccine with adjuvant — inactivated vaccine (vero cell) against EV71 of 400U /0.5ml, two doses, 28 days interval
  Other Names: EV71 vaccine
  Arms: 400U EV71 vaccine with adjuvant
Biological: 200U EV71 vaccine without adjuvant — inactivated vaccine (vero cell) against EV71 without adjuvant of 200U /0.5ml, two doses, 28 days interval
  Other Names: EV71 vaccine
  Arms: 200U EV71 vaccine without adjuvant
Biological: Placebo — 0.5ml placebo, two doses, 28 days interval
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, double-blind clinical trial is to evaluate the safety and immunogenicity of a new inactivated EV71 vaccine developed by Sinovac Biotech CO., LTD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, aged from 6 months to 11 years old Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
2. Provided legal identification for the sake of recruitment.
3. Subjects and/or parent(s)/legal guardian(s) are able to understand and sign informed consents.
4. Birth weight more than 2500 grams

Exclusion Criteria:

1. History of Hand-foot-mouth Disease
2. Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
3. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
4. Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
5. Epilepsy, seizures or convulsions history, or family history of mental illness
6. Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
7. History of asthma, angioedema, diabetes or malignancy
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
10. Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
11. Acute illness or acute exacerbation of chronic disease within the past 7 days
12. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
13. History of any blood products within 3 months
14. Administration of any live attenuated vaccine within 28 days
15. Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 14 days
16. Axillary temperature > 37.0 centigrade before vaccination
17. Abnormal laboratory parameters before vaccination
18. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Neutralization antibody geometric mean titer in infants 28 days after immunization with EV71 vaccine with or without aluminium hydroxide adjuvant | 6 month
  Primary immunogenicity end point were geometric mean titer of neutralization antibody againt EV71 virus >= 1:8

SECONDARY OUTCOMES:
The rates and severity of solicited adverse events in infants following immunization as a Measure of Safety and Tolerability | 6 months
  solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site.
  solicited general adverse events include Fever, Nausea, Vomiting, Diareahhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy

CONTACTS AND LOCATIONS:
Overall Officials: Yan-pin Li, MD, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- GuangXi Center for Diseases Control and Prevention, Nanning, Guangxi, China